CLINICAL TRIAL: NCT02891928
Title: Comparative Evaluation of Standard Wearing Shoes With Rocker Sole Shoes in Diabetic Patients With Neuropathy
Brief Title: Evaluation of Rocker sOles in Diabetis
Acronym: EROD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ROCKER SOLE (RB 14.143)
Record Dates: First submitted 2016-08-26; First posted 2016-09-08 (Estimated); Last update posted 2025-12-03 (Actual); Status verified 2016-09

CONDITIONS: Diabetic Neuropathy
Keywords: Type 2 diabetes; Diabetic neuropathy; Disorders of equilibrium; "Rocker sole" shoes; Walking
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- with rocker sole (Experimental): patient were wearing the rocker soles shoes during investigation
  Interventions: Device: Rocker sole shoes
- without rocker sole (Placebo Comparator): patient were wearing normal shoes during investigation
  Interventions: Device: Normal shoes

INTERVENTIONS:
Device: Rocker sole shoes — Measure of walk testing Measure of standing position
  Arms: with rocker sole
Device: Normal shoes — Measure of walk testing Measure of standing position
  Arms: without rocker sole

SUMMARY:
The purpose of this study is to determine if the wearing of shoes "rocker sole" type prescribed in type 2 diabetics patients with neuropathy are responsible for disorders of equilibrium.

DETAILED DESCRIPTION:
Diabetes is a public health problem. The functional prognosis is partly conditioned by the occurrence of wounds at the level of the foot affected by neuropathy and/or arteriopathy. Preventive measures are necessary to avoid such complications: education, pedicure, suitable footwear, insoles. There are many types of orthopedic shoes, standard or custom-made. A key objective is to avoid excessive pressure found at the level of the front-foot, favoring the appearance of lesions like ulcers. In this context, the Anglo-Saxons have developed a type of shoe ( "rocker sole"), allowing to decrease the pressures on the front-foot with a rigid sole system associated with an elevation of the front-foot. Some, however, have shown that this type of shoe may be responsible for disorders of equilibrium to the healthy subject, what about at the diabetic patients, already at higher risk of postural disorders and falls?

ELIGIBILITY:
Inclusion Criteria:

* Patient with Type 2 Diabetes
* Patients suffering from diabetic neuropathy diagnosed by the test in the monostrand
* Can walk without technical assistance
* Age from 18 to 75
* Having made his non-opposition

Exclusion Criteria:

* Presence of ulceration of the foot (or a history of this type)
* History of pathologies that could disturb the balance and walking independently of diabetes: vestibular diseases, ophthalmic diseases with decreased of visual acuity, neurological, musculoskeletal and rheumatic diseases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-12; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Anteroposterior displacement amount of the center of pressure with regard to the center of mass. | Inclusion
  Displacement of the center of pressure is measured during a 55 sec session of standing position with dedicated shoes with of force plateform

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Remy-Neris, Professor, Principal Investigator — CHRU de Brest
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: No
Data are not planned to be shared

REFERENCES:
- [Result] Lumeau M, Lempereur M, Remy-Neris O. Assessment of the rocker sole shoes on postural stability in diabetic patients with distal sensory neuropathy. Comput Methods Biomech Biomed Engin. 2015;18 Suppl 1:1986-7. doi: 10.1080/10255842.2015.1070588. Epub 2015 Aug 13. No abstract available. PMID 26269202